CLINICAL TRIAL: NCT01086527
Title: Genotype Stratified Pharmacokinetic Study of Montelukast
Acronym: GSPOM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Edward Mougey, Research Scientist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 37885; 32-03215-005 (Other: Nemours Children's Clinic)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Pharmacogenetics; Singulair; montelukast; Leukotriene Antagonists; Anti-Asthmatic Agents; Intestinal Absorption; pharmacokinetics; absorption; biochemical transport; Membrane Transport Proteins
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SLCO2B1{NM_007256.2}:c.[935G>A] + [=] (Experimental): Individuals in this group will be homozygous for SLCO2B1{NM_007256.2}:c.[935G>A].
  Interventions: Drug: 10 mg tablet of montelukast (Singulair)

INTERVENTIONS:
Drug: 10 mg tablet of montelukast (Singulair) — Fasting patients will take a single 10 mg tablet of montelukast with 240 ml of Gatorade. Eight blood samples will be drawn to assess the plasma concentration of montelukast over the subsequent 12 hours.
  Other Names: Singulair

SUMMARY:
Leukotriene receptor antagonists (LTRAs) are frequently prescribed to reduce the symptoms associated with asthma. Singulair (montelukast), manufactured by Merck, is a popular LTRA, however its effectiveness varies greatly between individuals. We are interested in understanding why the effectiveness of Singulair varies so greatly.

For an oral drug such as Singulair to be effective, the body must efficiently absorb it. We have found that blood levels of Singulair vary greatly between individuals, and we think that this variability is responsible for variability in response.

Drug absorption occurs primarily in the intestine. Due to differences in the chemical properties of drugs, some drugs can be absorbed easily while other drugs require help from special proteins produced by the cells that line the intestine. These proteins, or transporters act like revolving doors to allow drugs to move from the intestine to the bloodstream. The activity of a transporter can be influenced by individual genetic variability.

We think that adsorption of Singulair requires help from a transport protein called OATP2B1. We have found that a single common genetic change in this protein is associated with low plasma concentration of montelukast. In this proposal we will determine plasma levels of montelukast in individuals with two copies of this genetic change. We predict that these individuals will have roughly half the plasma level of montelukast as individuals with no copies of this genetic change.

Eventually, what we learn from this work will allow doctors to quickly test individuals with asthma to determine how well they will absorb Singulair and possibly other LTRAs. Knowing this will allow the doctor to adjust the drug treatment on an individual basis to maximize benefit in the treatment of asthma.

DETAILED DESCRIPTION:
We have previously reported that montelukast is a substrate for transport by OATP2B1 and that a common variant of SLCO2B1 (the gene coding for OATP2B1), c.[935G>A], which results in the substitution of Arg→Glu at amino acid position 312, was associated with steady-state plasma concentrations of montelukast and response(1). Compared to G/G homozygotes, A/G heterozygotes had lower plasma concentrations at both 1 and 6 months of therapy. Additionally, scores on the Asthma Symptom Utility Index were higher (better asthma control) in G/G homozygotes compared to A/G heterozygotes at both sampling intervals, but not prior to treatment. We concluded that genotype at c.935 may contribute to the variability in response to montelukast.

We recently completed a study of the influence of genotype at c.935 and the co-ingestion of citrus juice on the pharmacokinetics of a single 10-mg dose of montelukast in 26 adolescent subjects with physician-diagnosed asthma (NCT00513760). Twenty-one participants were genotyped as G/G homozygotes and five as A/G heterozygotes. The area under the montelukast plasma concentration vs. time curve (AUC) in A/G heterozygotes was 46% lower than the AUC in G/G homozygotes, replicating our earlier findings that genotype at c.935 influences the pharmacokinetics of montelukast.

Assuming an additive genetic model, our data predict that the AUC of montelukast in individuals carrying the A/A genotype would be even lower than in heterozygotes. The prevalence of the homozygous mutant allele (A/A) is low among African and European Americans (0 - 3%; http://www.ncbi.nlm.nih.gov/projects/SNP/). However the prevalence of the A/A genotype is 18% in both Asian Americans and Hispanics, and thus these racial / ethnic groups represent an ideal model to test the hypothesis that genotype at c.935 influences the pharmacokinetics and pharmacodynamics of montelukast. In this study, we will generate preliminary data showing that the AUC of montelukast is lowest in A/A, intermediate in A/G and highest in G/G and confirm the suitability of this model to replicate our earlier findings that genotype at c.935 is associated with response to montelukast.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be 7-35 years old.
* Individuals will be healthy or have doctor diagnosed asthma.
* Individuals 7-18 years old will have doctor diagnosed asthma.
* Individuals will have the (A/A) genotype at c.935.

Exclusion Criteria:

* Individuals must not be taking any oral medications except for ICS/or albuterol.
* Women must not be pregnant.

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2010-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC of montelukast | 0-12 hours
  Area under the concentration vs. time curve for the plasma concentration of montelukast.

SECONDARY OUTCOMES:
Ke of montelukast | 0-12 hours
  Elimination rate constant of montelukast.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Mougey, Ph.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Mougey EB, Feng H, Castro M, Irvin CG, Lima JJ. Absorption of montelukast is transporter mediated: a common variant of OATP2B1 is associated with reduced plasma concentrations and poor response. Pharmacogenet Genomics. 2009 Feb;19(2):129-38. doi: 10.1097/FPC.0b013e32831bd98c. PMID 19151602
- [Background] Mougey EB, Lang JE, Wen X, Lima JJ. Effect of citrus juice and SLCO2B1 genotype on the pharmacokinetics of montelukast. J Clin Pharmacol. 2011 May;51(5):751-60. doi: 10.1177/0091270010374472. Epub 2010 Oct 25. PMID 20974993